CLINICAL TRIAL: NCT00682084
Title: Insulin Sensitivity and Substrate Metabolism in Patients With Cushing's Syndrome Before and After Surgical Treatment
Brief Title: Insulin Sensitivity and Substrate Metabolism in Patients With Cushing's Syndrome
Status: Terminated | Type: Observational
Why Stopped: Recruitment problems
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MM-ISC-20070131
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2014-12

CONDITIONS: Cushing's Syndrome; Insulin Resistance
Keywords: Cushing's syndrome; Glucose tolerance; Insulin sensitivity; Substrate metabolism; Body composition
MeSH Terms: conditions — Cushing Syndrome; Insulin Resistance | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, muscle samples, fat samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients recently diagnosed with Cushing's syndrome
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgical removal of either a pituitary or ectopic ACTH producing tumor or an adrenal tumor

SUMMARY:
The purpose of this study is to investigate the effect og chronic elevated levels of cortisol on metabolism and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Age between 18 and 70
* Diagnosed with Cushing's syndrome

Exclusion Criteria:

* Suspected malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recently diagnosed with Cushing's syndrome, recruited from the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Before and after treatment

SECONDARY OUTCOMES:
Glucose tolerance, QoL, body composition, intrahepatic and intramyocellular fat, substrate metabolism. | Before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, Professor MD, Principal Investigator — Aarhus University Hospital, Department of Endocrinology
Locations (1):
- Department of Endocrinology, Aarhus C, Aarhus, Denmark